CLINICAL TRIAL: NCT01164475
Title: A Phase 4, Multicenter, Randomized, Comparator Trial Evaluating the Standard Weight-Based Dose (0.24 mg/kg) Compared to a Fixed Dose (20 mg) of Plerixafor Injection in Combination With G-CSF to Mobilize and Collect ≥5 x 10^6 CD34+ Cells/kg in ≤4 Days and to Evaluate the Difference in Total Systemic Exposure in Patients With Non-Hodgkin's Lymphoma Weighing ≤70 kg
Brief Title: Evaluation of Approved Weight-Based Dose Compared to Fixed Dose of Plerixafor in Patients With Non-Hodgkin's Lymphoma (NHL) Weighing Less Than 70 Kilograms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOZ11809; MSC12830 (Other: Other Company study code)
Record Dates: First submitted 2010-07-09; First posted 2010-07-16 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed Dose Plerixafor (Experimental): 10 microgram per kilogram (mcg/kg) granulocyte-colony stimulating factor (G-CSF) subcutaneous (SC) injection once daily in morning from Day 1 through Day 4 (G-CSF mobilization period), followed by 20 milligram (mg) plerixafor SC injection (fixed dose) in evening of Day 4 (10 to 11 hours prior to first apheresis), and then 10 mcg/kg G-CSF SC injection in morning of Day 5 (1 hour prior to first apheresis). Apheresis process and treatment with plerixafor (10 to 11 hours prior to apheresis) and G-CSF (1 hour prior to apheresis) was continued until the target number of cluster of differentiation 34 (CD34+) stem cells (greater than or equal to [>=] 5*10^6 cells/kg) was collected or until a maximum 4 apheresis sessions occurred.
  Interventions: Drug: Granulocyte-colony stimulating factor (G-CSF); Drug: Fixed Dose Plerixafor
- Weight-Based Plerixafor (Active Comparator): G-CSF 10 mcg/kg SC injection once daily in morning from Day 1 through Day 4 (G-CSF mobilization period), followed by plerixafor 0.24 milligram per kilogram (mg/kg) SC injection (weight-based dose) in evening of Day 4 (10 to 11 hours before first apheresis), and then G-CSF 10 mcg/kg SC injection in morning of Day 5 (1 hour prior to first apheresis). Apheresis process and treatment with plerixafor (10 to 11 hours prior to apheresis) and G-CSF (1 hour prior to apheresis) was continued until the target number of CD34+ stem cells (>=5*10^6 cells/kg) was collected or until a maximum 4 apheresis sessions occurred.
  Interventions: Drug: Granulocyte-colony stimulating factor (G-CSF); Drug: Weight-Based Plerixafor

INTERVENTIONS:
Drug: Granulocyte-colony stimulating factor (G-CSF)
  Other Names: Filgrastim
Drug: Fixed Dose Plerixafor
  Other Names: Mozobil; AMD3100
  Arms: Fixed Dose Plerixafor
Drug: Weight-Based Plerixafor
  Other Names: Mozobil; AMD3100
  Arms: Weight-Based Plerixafor

SUMMARY:
The purpose of this study was to compare the responses of 2 different doses of plerixafor in patients with Non-Hodgkin's Lymphoma (NHL) who received an autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 78 years (inclusive)
* Patients diagnosed with NHL who were to receive treatment with an autologous peripheral stem cell transplant for the first time
* Biopsy-confirmed diagnosis of NHL (chronic lymphocytic leukemia and all variants were excluded)
* Weight less than or equal to 70 kg
* In first or second complete remission or partial remission, defined for the purpose of this study as complete or partial response following first or second-line therapy only
* At least 4 weeks since last cycle of chemotherapy and/or other cancer therapy including rituximab
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Recovered from all acute toxic effects of prior chemotherapy
* Negative for human immunodeficiency virus (HIV), active hepatitis B, and active hepatitis C from assessments performed within 3 months before signing informed consent
* Signed informed consent form (ICF)
* White blood cell count (WBC) greater than (>) 2.5*10^9 per liter (L)
* Absolute neutrophil count (ANC) >1.5*10^9/L
* Platelet (PLT) count >100*10^9/L
* Creatinine clearance >=80 milliliter per minute (mL/min) (estimated by Cockcroft-Gault formula or 24 hour urine collection)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST), serum glutamic pyruvic transaminase (SGPT)/alanine aminotransferase (ALT), and total bilirubin less than 2.5*upper limit of normal
* Cardiac and pulmonary status sufficient to undergo apheresis and transplantation
* All patients agreed to an effective method of contraception while on study treatment and for at least 3 months following plerixafor treatment (including both female patients of child-bearing potential and male patients with partners of child-bearing potential)

Exclusion Criteria:

* A co-morbid condition which, in the view of the Investigator(s), rendered the patient at high risk from treatment complications
* Failed previous hematopoietic stem cell (HSC) collections or collection attempts
* Prior autologous or allogeneic transplant
* Less than 6 weeks off 1,3-bis (2-chloroethyl)-1-nitroso-urea (BCNU) prior to first dose of G-CSF
* Active central nervous system involvement, active brain metastases, or any history of carcinomatous meningitis (active or inactive)
* Bone marrow involvement >20 percent (%), as assessed by bone marrow biopsy within 4 months of the first screening assessment, unless a bone marrow biopsy was performed immediately prior to the last chemotherapy and was negative and the patient responded to last chemotherapy achieving a complete or partial remission
* Received radiation therapy to the pelvis
* Received granulocyte/macrophage-colony stimulating factor (GM-CSF) or pegfilgrastim within 3 weeks prior to the first dose of granulocyte colony stimulating factor (G-CSF) for mobilization
* Received G-CSF within 14 days prior to the first dose of G-CSF for mobilization
* Received prior radio-immunotherapy with ibritumomab tiuxetan or tositumomab iodine
* Active infection, including unexplained fever (>38.1 degree Celsius / 100.4 Fahrenheit), or antibiotic, antiviral, or antifungal therapy within 7 days prior to the first dose of G-CSF
* Positive pregnancy test (female patients)
* Lactating (female patients)
* Abnormal electrocardiogram (ECG) with clinically significant rhythm disturbance (ventricular arrhythmias) or other conduction abnormality in the last year that, in the opinion of the Investigator(s), warranted exclusion of the patient from the trial
* Previously received experimental therapy within 4 weeks of enrolling or who were currently enrolled in another experimental protocol during the G CSF and plerixafor treatment period

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- United States (2):
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Cancer Center, Aurora, Colorado
- Princess Margaret Hospital, Toronto, Ontario, Canada
- South Korea (2):
  - Samsung Medical Center, Seoul
  - St. Mary's Hospital, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers in 4 countries between October 13, 2010 and February 26, 2013.
Pre-assignment Details: A total of 71 patients were screened of which 10 patients were screen failures. A total of 61 patients were randomized.
Period: Overall Study
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Started | 30 | 31
Completed | 28 | 29
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other | 0 | 1
Not completed — Progressive disease | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Groups:
- Fixed Dose Plerixafor: 10 microgram per kilogram (mcg/kg) granulocyte-colony stimulating factor (G-CSF) subcutaneous (SC) injection once daily in morning from Day 1 through Day 4 (G-CSF mobilization period), followed by 20 milligram (mg) plerixafor SC injection (fixed dose) in evening of Day 4 (10 to 11 hours prior to first apheresis), and then 10 mcg/kg G-CSF SC injection in morning of Day 5 (1 hour prior to first apheresis). Apheresis process and treatment with plerixafor (10 to 11 hours prior to apheresis) and G-CSF (1 hour prior to apheresis) was continued until the target number of cluster of differentiation 34 (CD34+) stem cells (>=5*10^6 cells/kg) was collected or until a maximum 4 apheresis sessions occurred.
- Total: Total of all reporting groups
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.13 (13.40) | 47.84 (13.59) | 47.00 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 12 | 14 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Asian | 28 | 28 | 56
  Race: White | 2 | 3 | 5
  Ethnicity: Hispanic or Latino | 1 | 2 | 3
  Ethnicity: Not Hispanic or Latino | 29 | 29 | 58
Number of Patients With Peripheral-Blood (PB) Cluster of Differentiation 34+ (CD34+) Cell Count [Number; unit: participants] — Baseline for this characteristic was "pre G-CSF dose on Day 4"
  participants
    Less than 10 cells per microliter (mcL) | 20 | 21 | 41
    Greater than or equal to 10 cells/mcL | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieved at Least 5*10^6 Cluster of Differentiation 34+ (CD34+) Cells Per Kilogram (Cells/kg)
Description: The cumulative number of CD34+ cells/kg (body weight) collected over all apheresis sessions (up to a maximum of 4 sessions) was used to determine if a patient has achieved the target of >=5*10^6 CD34+ cells/kg (optimum number of CD34+ cells required for transplantation) within 4 days of apheresis. The proportion of patients who achieved the target was reported as percentages for each treatment arm.
Time Frame: Day 5 up to Day 8
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Number; unit: percentage of participants
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
percentage of participants | 60.0 | 54.8
Statistical Analysis 1: Comparison: Fixed Dose Plerixafor vs Weight-Based Plerixafor; The comparison was done using the logistic regression model, adjusted for country and baseline PB CD34+ cell count; Test type: Superiority or Other; p = 0.395, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.44 to 9.17]

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 10 Hours (AUC [0-10])
Time Frame: 0 (pre-plerixafor dose), 0.5, 1, 4 hours post-plerixafor dose on Day 4; 9-10 hours post-plerixafor dose (pre G-CSF dose) on Day 5, 10-11 hours post-plerixafor dose (prior to first apheresis) on Day 5
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Geometric Mean (Standard Error); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
nanogram*hour per milliliter (ng*hr/mL) | 3991.2 (1.03) | 2792.7 (1.03)

3. Secondary Outcome: Proportion of Patients Who Achieved at Least 2*10^6 CD34+ Cells/kg in Less Than or Equal to 4 Days of Apheresis
Description: The cumulative number of CD34+ cells/kg (body weight) collected over all apheresis sessions (up to a maximum of 4 sessions) was used to determine if a patient has achieved the target of >= 2*10^6 CD34+ cells/kg (minimum number of CD34+ cells required for transplantation) within 4 days of apheresis. The proportion of patients who achieved the target was reported as percentages for each treatment arm.
Time Frame: Day 5 up to Day 8
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Number; unit: percentage of participants
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
percentage of participants | 93.3 | 90.3

4. Secondary Outcome: Median Number of Days of Apheresis to Collect at Least 2*10^6 CD34+ Cells/kg
Time Frame: Day 5 up to Day 8
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor. Here, number of patients analyzed = the number of patients who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 28 | 28
days | 1 [1 to 4] | 2 [1 to 4]

5. Secondary Outcome: Median Number of Days of Apheresis to Collect at Least 5*10^6 CD34+ Cells/kg
Time Frame: Day 5 up to Day 8
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 18 | 17
days | 3 [1 to 4] | 3 [1 to 4]

6. Secondary Outcome: Total Number of CD34+ Cells/kg Collected Over up to 4 Aphereses
Description: The cumulative number of CD34+ cells/kg (body weight) collected over all apheresis sessions (up to a maximum of 4 sessions) was reported.
Time Frame: Day 5 up to Day 8
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Median (Full Range); unit: 10^6 cells/kg
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
10^6 cells/kg | 5.35 [1.2 to 9.6] | 5.24 [1.3 to 372.8]

7. Secondary Outcome: Mean Fold Increase in Peripheral Blood CD34+ Cell Count Following Plerixafor
Description: Fold increase was calculated as CD34+ cell count on Day 5 divided by CD34+ cell count on Day 4.
Time Frame: Baseline (pre G-CSF dose on Day 4) to Day 5 (prior to first apheresis)
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Mean (Standard Deviation); unit: fold increase
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
fold increase | 5.43 (4.02) | 5.09 (2.81)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
ng/mL | 957 (216) | 711 (136)

9. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Population: FAS included all patients who have signed informed consent and received at least one dose of study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
hours | 0.50 [0.42 to 1.08] | 0.50 [0.42 to 1.02]

10. Secondary Outcome: Terminal Elimination Half-life (T1/2)
Description: T1/2 is the time required for the plasma concentration to decrease to one half.
Time Frame: as for outcome 2
Population: FAS included all randomized patients who signed informed consent form and received at least one dose of plerixafor.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Number analyzed (Participants) | 30 | 31
hours | 4.53 (1.38) | 4.27 (0.93)

ADVERSE EVENTS:
Time Frame: From signing of inform consent form up to 30 days after the last dose of plerixafor
Description: Median number of plerixafor doses was 3 doses for both treatment arms. The analysis was performed on safety population, defined as all patients who signed informed consent form and received at least one dose of plerixafor.
Arm/Group | Fixed Dose Plerixafor | Weight-Based Plerixafor
Serious Adverse Events (participants affected / at risk) | 0/30 | 3/31
Other Adverse Events (participants affected / at risk) | 26/30 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Dose Plerixafor (N=30) | Weight-Based Plerixafor (N=31)
Cellulitis (Infections and infestations) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Dose Plerixafor (N=30) | Weight-Based Plerixafor (N=31)
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 7
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 4 | 2
Catheter site pain (General disorders) | 1 | 2
Chest discomfort (General disorders) | 2 | 0
Injection site erythema (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 3 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 2
Blood calcium decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 3
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 4 | 3
Lymphocyte percentage decreased (Investigations) | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 0
Monocyte count increased (Investigations) | 2 | 2
Neutrophil count increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 14 | 8
Protein total (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 1
Red blood cell count decreased (Investigations) | 2 | 1
Red cell distribution width increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Fluid overload (Metabolism and nutrition disorders) | 3 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Anaesthesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 2
Monoplegia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.